CLINICAL TRIAL: NCT06147908
Title: A Bioequivalence Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety After Administration of DW5221 and DW5221-R in Healthy Adult Male Volunteers
Brief Title: Clinical Trial to Evaluate the Pharmacokinetic Characteristics of DW5221 and DW5221-R
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW5221-1
Record Dates: First submitted 2023-11-15; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Apetite Stimulants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): cross-over
  Interventions: Drug: DW5221; Drug: DW5221-R
- Sequence B (Experimental): cross-over
  Interventions: Drug: DW5221; Drug: DW5221-R

INTERVENTIONS:
Drug: DW5221 — megestrol acetate
  Other Names: Test
Drug: DW5221-R — megestrol acetate
  Other Names: Reference

SUMMARY:
A bioequivalence study to compare and evaluate the pharmacokinetic characteristics and the safety after administration of DW5221 and DW5221-R in healthy adult m ale volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male Volunteers who are ≥19 years old
* Body weight ≥50.0 kg and BMI between 18.0 and 30.0 kg/m2 and

Exclusion Criteria:

* Clinically significant Medical History

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 120 hour
  Pharmacokinetics of Megestrol Acetate
Area under the plasma concentration versus time curve (AUC) | up to 120 hour
  Pharmacokinetics of Megestrol Acetate

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

REFERENCES:
- [Derived] Park SR, Hwang JG, Jeong SI, Choi YS, Min HJ, Kim HY, Choi BH, Park MK. Comparison of the pharmacokinetic characteristics and bioequivalence between two nanosuspension formulations of megestrol acetate in healthy Korean male subjects. Transl Clin Pharmacol. 2024 Mar;32(1):63-72. doi: 10.12793/tcp.2024.32.e6. Epub 2024 Mar 26. PMID 38586120